CLINICAL TRIAL: NCT03634267
Title: MRI Guided Brachytherapy for HPV-Associated Cervical and Vaginal Malignancies
Brief Title: MRI-Guided Brachytherapy in Treating Participants With HPV-Associated Stage IB2-IVA Cervical or Stage II-IVA Vaginal Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-0823; NCI-2018-01569 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-0823 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2018-08-03; First posted 2018-08-16 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Human Papillomavirus-Related Carcinoma; Human Papillomavirus-Related Cervical Carcinoma; Stage IB2 Cervical Cancer AJCC v8; Stage II Cervical Cancer AJCC v8; Stage II Vaginal Cancer AJCC v8; Stage IIA Cervical Cancer AJCC v8; Stage IIA Vaginal Cancer AJCC v8; Stage IIA1 Cervical Cancer AJCC v8; Stage IIA2 Cervical Cancer AJCC v8; Stage IIB Cervical Cancer AJCC v8; Stage IIB Vaginal Cancer AJCC v8; Stage III Cervical Cancer AJCC v8; Stage III Vaginal Cancer AJCC v8; Stage IIIA Cervical Cancer AJCC v8; Stage IIIB Cervical Cancer AJCC v8; Stage IVA Cervical Cancer AJCC v8; Stage IVA Vaginal Cancer AJCC v8
MeSH Terms: conditions — Uterine Cervical Neoplasms; Vaginal Neoplasms | interventions — Brachytherapy; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (MRI, internal radiation therapy) (Experimental): Participants undergo MRI scan during internal radiation therapy applicator placement.
  Interventions: Radiation: Internal Radiation Therapy; Procedure: Magnetic Resonance Imaging

INTERVENTIONS:
Radiation: Internal Radiation Therapy — Undergo brachytherapy
  Other Names: BRACHYTHERAPY; internal radiation; Internal Radiation Brachytherapy; Radiation Brachytherapy
Procedure: Magnetic Resonance Imaging — Undergo MRI scan
  Other Names: Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging

SUMMARY:
This trial studies how well magnetic resonance imaging (MRI)-guided internal radiation therapy (brachytherapy) works in treating participants with human papillomavirus (HPV) associated stage IB2-IV cervical or stage II-IVA vaginal cancer. Using MRI guidance during brachytherapy applicator placement may improve treatment planning in participants with cervical or vaginal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine whether MRI guidance during internal radiation therapy applicator placement improves the high-risk clinical target volume (HR-CTV) D90 (dose to 90% of the high-risk clinical target volume) rate compared to conventional guidance, with ultrasound and freehand technique, for patients with cervical and vaginal cancer.

SECONDARY OBJECTIVES:

I. Identify diffusion weighted MRI image features that can be used to identify sites of viable tumor following external beam radiotherapy as assessed by tumor aspirate cytology.

II. Determine if diffusion weighted MRI findings are associated with immune infiltration as assessed by multi-spectral flow cytometry.

III. Identify potential correlates between clinical outcomes (survival, progression) and these data objectives (brachytherapy dosimetry/therapeutic ratio, diffusion-weighted MRI imaging features, tumor aspirate cytology findings).

IV. Define the financial costs and feasibility of an MRI-guided brachytherapy approach to determine the overall healthcare quality value (outcomes/cost) of this novel approach for application at other brachytherapy centers.

OUTLINE:

Participants undergo MRI scan during internal radiation therapy applicator placement.

ELIGIBILITY:
Inclusion Criteria:

* Women with stage 1B2-IVA cervical cancer recommended to receive definitive chemoradiation including brachytherapy; or
* Women with stage II-IVA vaginal cancer recommended to receive definitive chemoradiation including brachytherapy.

Exclusion Criteria:

* Patient or tumor anatomy that requires use of a non-MRI-compatible applicator.
* Patients with implantable cardioverter-defibrillator, pacemaker or other implanted device or medical condition which precludes MRI acquisition.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-08-03 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Percent of patients achieving high-risk clinical target volume (HR-CTV) dose to 90% (D90) | Up to 4 years
  Rate will be compared to conventional guidance, with ultrasound and freehand technique. We will compare the HR-CTV D90 and other secondary dosimetry parameters (e.g. D2 cc bladder, D2 cc rectum etc.) between the initial scan (subsequent to ultrasound [US] guided or freehand applicator placement) and optimized (with magnetic resonance imaging [MRI] guided placement) treatment plan for each patient using McNemar's test.

SECONDARY OUTCOMES:
Diffusion weighted imaging (DWI) outcomes | Up to 4 years
Biomarker measurements (tumor viability and tumor T cell profile) from tumor samples | Up to 4 years
  A paired t-test will be used to compare apparent diffusion coefficient (ADC) areas for each biomarker.
Disease recurrence (local, regional, and distant) | Up to 4 years
  determined via axial imaging (MRI or PET/CT) on interval follow-up
Overall survival | Up to 4 years
Progression-free survival | Up to 4 years
Incidence and severity of treatment-related toxicities | Up to 4 years
  as defined via CTCAE v4.0
Cost difference associated with the MRI-guided versus the standard process | Up to 4 years
  Billing and financial data will be calculated and compared to that of the conventional non-MRI-guided brachytherapy approach.

CONTACTS AND LOCATIONS:
Overall Officials: Ann H Klopp, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org